CLINICAL TRIAL: NCT01311557
Title: Safety and Immunogenicity of Adacel® Vaccine Administered to Persons 10 Years of Age
Brief Title: Study of Adacel® Vaccine Administered to Persons 10 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Td519; U1111-1115-6619 (Other: WHO)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Tetanus; Diphtheria; Pertussis
Keywords: Tetanus; Diphtheria; Pertussis; Tdap vaccine; Adacel®
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adacel Vaccine Group 1 (Experimental): Participants enrolled at 10 to < 11 years of age
  Interventions: Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Adsorbed
- Adacel Vaccine Group 2 (Experimental): Participants enrolled at 11 to < 12 years of age
  Interventions: Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Adsorbed

INTERVENTIONS:
Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Adsorbed — 0.5 mL, Intramuscular
  Other Names: Adacel®
  Arms: Adacel Vaccine Group 1
Biological: Adacel®: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Adsorbed — 0.5 mL, Intramuscular
  Other Names: Adacel®
  Arms: Adacel Vaccine Group 2

SUMMARY:
The purpose of study Td519 is to demonstrate that Adacel® vaccine (Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Adsorbed) is safe and immunogenic in persons 10 years of age.

Primary Objectives:

* To compare pertussis antibody responses induced by Adacel® in persons 10 to <11 years of age to those induced by Adacel in persons 11 to <12 years of age.
* To compare the booster responses against pertussis antigens induced by Adacel in persons 10 to <11 years of age to those induced by Adacel in persons 11 to <12 years of age.
* To compare booster responses against tetanus and diphtheria induced by Adacel in persons 10 to <11 years of age to those induced by Adacel in persons 11 to <12 years of age.

Secondary Objective:

* To compare seroprotection rates against tetanus and diphtheria induced by Adacel in persons 10 to <11 years of age to those induced by Adacel in persons 11 to <12 years of age.

DETAILED DESCRIPTION:
Study participants will receive a single dose of study vaccine and will then be monitored for safety from the day of vaccination for up to 30 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age is > 10 to < 12 years of age at the time of vaccination.
* Assent form has been signed and dated by the subject, and informed consent has been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures.
* For a female of childbearing potential, abstinence or use of an effective method of contraception from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.
* Documented vaccination history of receiving 5 previous doses of DTaP (combination diphtheria, tetanus, and acellular pertussis) vaccine (consisting of 3 infant doses in the first year of life, a 4th dose in the 2nd year of life, and a 5th dose at 4 through 6 years of age).

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Serious, acute, or chronic disease that is unstable or that, in the opinion of the Investigator, might: (i) interfere with the ability to participate fully in the study; or (ii) interfere with evaluation of the vaccine.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Prior receipt of pertussis, diphtheria, or tetanus containing vaccines within the past 5 years.
* A personal history of physician-diagnosed or laboratory confirmed pertussis disease within the last 2 years.
* A previous severe reaction to pertussis, diphtheria or tetanus vaccine including immediate anaphylaxis, encephalopathy within 7 days or seizure within 3 days of receiving the vaccine.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with the assessment of the immune response.
* History of allergy to egg proteins, latex, or any constituents of the vaccine.
* Suspected or known hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before the 2nd visit; except that influenza vaccine may have been received between 30 and 15 days (but no less than 15 days) before receiving study vaccine.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study.
* Seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, as reported by the parent/guardian.
* Laboratory-confirmed thrombocytopenia, bleeding disorders, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination, at the discretion of the Investigator.
* Known pregnancy, or a positive urine or serum pregnancy test.
* Prior personal history of Guillain-Barré syndrome.
* Identified as an investigator or employee of the investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the investigator or employee with direct involvement in the proposed study.

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1302 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (34):
- United States (34):
  - Chandler, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Sacramento, California
  - Longmont, Colorado
  - Norwich, Connecticut
  - Miami Beach, Florida
  - Marietta, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Haughton, Louisiana
  - Metairie, Louisiana
  - Woburn, Massachusetts
  - Plymouth, Minnesota
  - Rochester, New York
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Barnwell, South Carolina
  - Rapid City, South Dakota
  - Kingsport, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Midlothian, Virginia
  - Vienna, Virginia
  - Spokane, Washington
  - Marshfield, Wisconsin

REFERENCES:
- [Derived] Marshall GS, Pool V, Greenberg DP, Johnson DR, Sheng X, Decker MD. Safety and immunogenicity of tetanus-diphtheria-acellular pertussis vaccine administered to children 10 or 11 years of age. Clin Vaccine Immunol. 2014 Nov;21(11):1560-4. doi: 10.1128/CVI.00474-14. Epub 2014 Sep 17. PMID 25230939
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 07 March 2011 to 19 May 2011 at 36 clinical centers in the United States.
Pre-assignment Details: A total of 1302 participants who met all inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Participants 10 to <11 Years of Age; Participants 11 to <12 Years of Age: Participants received 1 dose of Adacel® vaccine at Visit 1.
Period: Overall Study
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Started | 651 | 651
Completed | 646 | 645
Not Completed | 5 | 6
Not completed — Serious adverse event | 0 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age | Total
Number analyzed (Participants) | 651 | 651 | 1302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 651 | 651 | 1302
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.5 (0.3) | 11.4 (0.3) | 10.5 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 315 | 620
  Male | 346 | 336 | 682
Region of Enrollment [Number; unit: Participants]
  United States | 651 | 651 | 1302

OUTCOME MEASURES:

1. Primary Outcome: Summary of Geometric Mean Titers of Anti-Pertussis Titers Following a Single Dose of Adacel® Vaccine
Description: Anti-Pertussis titers (Pertussis toxoid [PT], Filamentous hemagglutinin [FHA], Pertactin [PRN], Fimbriae types 2 and 3 [FIM]) geometric mean titers were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 30 post-vaccination
Population: Geometric mean titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 613 | 608
Titers (1/dilutions)
  Anti-Pertussis toxoid (N=577, 566) | 30.1 [28.0 to 32.4] | 32.0 [29.6 to 34.7]
  Anti-Filamentous hemagglutinin, Day 30(N=613, 608) | 232 [218 to 247] | 225 [211 to 239]
  Anti-Pertactin (N=613, 607) | 464 [426 to 506] | 444 [408 to 482]
  Anti-Fimbriae types 2 & 3 (N=606, 605) | 477 [413 to 550] | 540 [478 to 611]
Statistical Analysis 1: Comparison: Participants 10 to <11 Years of Age vs Participants 11 to <12 Years of Age; Test type: Non-Inferiority or Equivalence — A two-sided 95% confidence interval (CI) was constructed around each of the ratios: Pertussis toxoid (PT) GMT Group 1 / GMT Group 2. The GMT hypothesis was supported by the data if the lower bound of the calculated 95% CI was > 0.67. This was the equivalent of testing the null hypothesis using a one-sided type I error rate of 0.025; GMT Ratio = 0.940, 95% CI 2-sided [0.843 to 1.05]
Statistical Analysis 2: Comparison: Participants 10 to <11 Years of Age vs Participants 11 to <12 Years of Age; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was constructed around each of the ratios: anti-Filamentous hemagglutinin (FHA) GMT Group 1 / GMT Group 2. The GMT hypothesis was supported by the data if the lower bound of the calculated 95% CI was > 0.67. This was the equivalent of testing the null hypothesis using a one-sided type I error rate of 0.025; GMT Ratio = 1.03, 95% CI 2-sided [0.944 to 1.13]
Statistical Analysis 3: Comparison: Participants 10 to <11 Years of Age vs Participants 11 to <12 Years of Age; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was constructed around each of the ratios: Anti-Pertactin (PRN) GMT Group 1 / GMT Group 2. The GMT hypothesis was supported by the data if the lower bound of the calculated 95% CI was > 0.67. This was the equivalent of testing the null hypothesis using a one-sided type I error rate of 0.025; GMT Ratio = 1.05, 95% CI 2-sided [0.928 to 1.18]
Statistical Analysis 4: Comparison: Participants 10 to <11 Years of Age vs Participants 11 to <12 Years of Age; Test type: Non-Inferiority or Equivalence — A two-sided 95% CI was constructed around each of the ratios: anti-Fimbriae types 2 and 3 (FIM) GMT Group 1 / GMT Group 2. The GMT hypothesis was supported by the data if the lower bound of the calculated 95% CI was > 0.67. This was the equivalent of testing the null hypothesis using a one-sided type I error rate of 0.025; GMT Ratio = 0.882, 95% CI 2-sided [0.731 to 1.06]

2. Primary Outcome: Summary of Anti-Pertussis Booster Response Following a Booster Dose of Adacel® Vaccine
Description: Anti-Pertussis booster responses were assessed by enzyme linked immunosorbent assay (ELISA). For pertussis antigens (Pertussis toxoid [PT], filamentous hemagglutinin [FHA], pertactin [PRN], fimbriae types 2 and 3 [FIM]), a booster response rate was defined as a four-fold increase in pre- to post-vaccination titers for participants with pre vaccination titers ≤ 93 ELISA Unit (EU)/mL for PT, ≤ 170 EU/mL for FHA, ≤ 115 EU mL for PRN, and ≤ 285 EU/mL for FIM. If the pre-vaccination titers were > 93 EU/mL for PT, > 170 EU/mL for FHA, > 115 EU mL for PRN, or > 285 EU/mL for FIM then a two-fold increase in the antibody titer was defined as a booster response.
Time Frame: 30 days post-vaccination
Population: Anti-pertussis booster response were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 613 | 608
Percentage of participants
  Anti-Pertussis toxoid (N=554, 549) | 56.7 | 56.1
  Anti-filamentous hemagglutinin (N=609, 605) | 84.2 | 84.8
  Anti-Pertactin (N=600, 600) | 98.0 | 97.5
  Anti-Fimbriae types 2 and 3 (N=583, 585) | 93.7 | 97.1

3. Primary Outcome: Summary of Anti-Tetanus and Anti-Diphtheria Booster Response Following a Booster Dose of Adacel® Vaccine
Description: Anti-tetanus booster responses were assessed by enzyme-linked immunosorbent assay (ELISA). Anti-diphtheria booster responses were assessed by a toxin neutralization test. Booster response rate was defined as a four-fold increase in pre- to post-vaccination for subjects with pre-vaccination titers ≤ 2.56 EU/mL for diphtheria and ≤ 2.7 EU/mL for tetanus. If the pre-vaccination titers were > 2.56 EU/mL for diphtheria or > 2.7 EU/mL for tetanus, then a two-fold increase in response rate was defined as a booster response.
Time Frame: 30 days post-vaccination
Population: Anti-Tetanus and anti-Diphtheria booster responses were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 613 | 608
Percentage of participants
  Anti-Tetanus (N=610, 603) | 98.5 | 98.8
  Anti-Diphtheria (N=609, 605) | 97.7 | 98.0

4. Secondary Outcome: Percentage of Participants With Seroprotection to Tetanus and Diphtheria Following a Single Dose of Adacel Vaccine
Description: Anti-tetanus seroprotection rates were assessed by enzyme-linked immunosorbent assay (ELISA). Anti-diphtheria seroprotection was assessed by a toxin neutralization test. Seroprotection was defined as post-vaccination antibody titers ≥0.1 IU/mL.
Time Frame: Day 0 (pre-vaccination) and 30 days post-vaccination
Population: Seroprotection rates were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 613 | 608
Percentage of participants
  Anti-Tetanus (Pre-vaccination, N=610, 604) | 90.3 | 91.2
  Anti-Tetanus (Post-vaccination, N=613, 607) | 99.7 | 100.0
  Anti-Diphtheria (Pre-vaccination, N=610, 605) | 83.6 | 75.9
  Anti-Diphtheria (Post-vaccination, N=612, 608) | 99.7 | 100.0

5. Secondary Outcome: Summary of Anti-Pertussis Geometric Means of Titers Before and Post-Vaccination With a Single Dose of Adacel Vaccine
Description: Anti-Pertussis titers (Pertussis toxoid [PT], Filamentous hemagglutinin [FHA], Pertactin [PRN], Fimbriae types 2 and 3 [FIM]) geometric mean titers were assessed by enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 613 | 608
Titers (1/dilutions)
  Anti-Pertussis toxoid; Day 0 (N = 590, 591) | 4.96 [4.54 to 5.42] | 4.85 [4.41 to 5.34]
  Anti-Pertussis toxoid; Day 30 (N = 577, 566) | 30.1 [28.0 to 32.4] | 32.0 [29.6 to 34.7]
  Anti-Filamentous hemagglutinin Day 0 (N=609, 605) | 22.1 [20.1 to 24.2] | 20.3 [18.5 to 22.3]
  Anti-Filamentous hemagglutinin Day 30 (N=613, 608) | 232 [218 to 247] | 225 [211 to 239]
  Anti-Pertactin; Day 0 (N = 600, 601) | 15.6 [14.2 to 17.1] | 14.8 [13.5 to 16.2]
  Anti-Pertactin; Day 30 (N = 613, 607) | 464 [426 to 506] | 444 [408 to 482]
  Anti-Fimbriae types 2 and 3; Day 0 (N = 590, 587) | 6.77 [6.05 to 7.57] | 7.07 [6.33 to 7.89]
  Anti-Fimbriae types 2 and 3; Day 30 (N = 606, 605) | 477 [413 to 550] | 540 [478 to 611]

6. Secondary Outcome: Percentage of Participants Reporting a Solicited Injection-site or Systemic Reactions Following Injection With a Single Dose of Adacel Vaccine
Description: Solicited injection-site: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, and Myalgia. Grade 3 Solicited Injection-site reactions: Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, ≥50 mm. Grade 3 Solicited systemic reactions: Fever, ≥39.0˚C or ≥102.1˚F; Headache, Malaise, and Myalgia Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Number analyzed (Participants) | 650 | 649
Percentage of participants
  Injection-site Pain (N=644, 645) | 80.9 | 80.9
  Grade 3 Injection-site Pain (N=644, 645) | 3.3 | 2.2
  Injection-site Erythema (N=644, 645) | 39.4 | 38.4
  Grade 3 Injection-site Erythema (N=644, 645) | 7.9 | 7.4
  Injection-site Swelling (N=644, 645) | 35.2 | 33.5
  Grade 3 Injection-site Swelling (N=644, 645) | 8.4 | 7.3
  Fever (N=642, 644) | 1.6 | 0.6
  Grade 3 Fever (N=642, 644) | 0 | 0.2
  Headache (N=644, 646) | 33.1 | 37.6
  Grade 3 Headache (N=644, 646) | 2.0 | 1.9
  Malaise (N=644, 646) | 26.2 | 29.3
  Grade 3 Malaise (N=644, 646) | 1.9 | 2.8
  Myalgia (N=644, 645) | 49.1 | 56.4
  Grade 3 Myalgia (N=644, 645) | 3.3 | 1.7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 30 post-vaccination
Description: Solicited (non serious) adverse events were recorded in diary cards by the study participants or their guardians within 7 days after vaccination.
Arm/Group | Participants 10 to <11 Years of Age | Participants 11 to <12 Years of Age
Serious Adverse Events (participants affected / at risk) | 0/651 | 1/651
Other Adverse Events (participants affected / at risk) | 521/651 | 522/651
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants 10 to <11 Years of Age (N=651) | Participants 11 to <12 Years of Age (N=651)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants 10 to <11 Years of Age (N=651) | Participants 11 to <12 Years of Age (N=651)
Injection-site Pain (General disorders) | 521 (521) | 522 (522)
Injection-site Erythema (General disorders) | 254 (254) | 248 (248)
Injection-site Swelling (General disorders) | 227 (227) | 216 (216)
Headache (Nervous system disorders) | 213 (213) | 243 (243)
Malaise (General disorders) | 169 (169) | 189 (189)
Myalgia (Musculoskeletal and connective tissue disorders) | 316 (316) | 364 (364)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications